CLINICAL TRIAL: NCT01428232
Title: Comparison of Two Clinic-based Interventions to Promote Early Initiation and Exclusive Breastfeeding Through 6 Months After Birth in Kinshasa, Democratic Republic of Congo
Brief Title: Effectiveness of Well-child Clinics as the "Community" Basis of Step 10 of the Baby Friendly Hospital Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kinshasa School of Public Health (DR, Congo) (Unknown); Centre for the Coordination of Social Science Research and Documentation in Africa South of the Sahara (CERDAS) (DR,Congo) (Unknown); Bureau Diocésain des Œuvres Médicales de Kinshasa (BDOM), (DR, Congo) (Unknown); Salvation Army (DR, Congo) (Unknown); Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09-000076-AT11-123-UNC-DRC
Record Dates: First submitted 2011-08-29; First posted 2011-09-02 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-01

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Baby Friendly Hospital Initiative; Well-child clinics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BFHI steps 1-9 (Experimental): Hospital retrained in BFHI steps 1-9 Mothers can call hospital to obtain BF support/Mothers given phone # of maternity nurse whom she can call or go see if she has BF problems
  Interventions: Other: implementation of the Baby-Friendly Hospital Initiative
- BFHI steps 1-9 +well-child clinic (Experimental): Hospital retrained in BFHI steps 1-9 Mothers can call hospital to obtain BF support/Mothers given phone # of maternity nurse whom she can call or go see if she has BF problems Provision of BF support during 1) clinic visit to obtain birth certificate or home visit if mother does not come into clinic and 2) well-child clinics Flyers to mother with culturally appropriate messages designed to address some of the most important local barrier to EBF
  Interventions: Other: BFHI steps 1-9 +well-child clinic
- usual care (No Intervention)

INTERVENTIONS:
Other: implementation of the Baby-Friendly Hospital Initiative — Implementation of BFHI steps 1-9 in maternities
  Arms: BFHI steps 1-9
Other: BFHI steps 1-9 +well-child clinic — Implementation of BFHI steps 1-9 in maternities and provision of breastfeeding support including culturally appropriate educational messages and metaphors as the ongoing aspect of step 10 in well-child clinic
  Arms: BFHI steps 1-9 +well-child clinic

SUMMARY:
A cluster-randomized controlled trial will be conducted in the Democratic Republic of Congo to compare rates of early initiation and exclusive breastfeeding between mothers who give birth in hospitals with the current standard of care, mothers who give birth in hospitals that have implemented the first nine steps of the Baby-Friendly Hospital Initiative, and mothers who give birth in hospitals that have implemented all ten steps of the Baby-Friendly Hospital Initiative, with the 10th step being the provision of breastfeeding support during well-child clinic visits.

DETAILED DESCRIPTION:
If at least 90% of children were exclusively breastfed for the first 6-months of life, the potential reduction in mortality that can be achieved will be higher than for any other interventions with sufficient evidence of effect. In the DRC >500,000 under-five deaths occurred in 2008. While >95% of children were breastfed at some point, 18% received something other than breast milk before initiation of breastfeeding, and half received something other than human milk by 1.4 months. Pre- and post-partum breastfeeding support has been shown to best improve the rate of exclusive breastfeeding (EBF). The global initiatives to improve breastfeeding practices have focused on maternity-level policies and procedures known as the Ten Steps to Successful Breastfeeding, which served as the basis for the Baby-Friendly Hospital Initiative. These quality of care steps impact hospital breastfeeding rates as well as breastfeeding rates throughout the 6 months postpartum period. However, EBF rates fall off rapidly in the DRC. In the proposed cluster randomized controlled trial, we plan to evaluate the effect of breastfeeding support provided by well-child clinic staff including the use of culturally appropriate messages in addition to the implementation of BFHI steps 1-9 Steps in maternities on the rate of breastfeeding initiation within 1 hour of birth and EBF throughout 6 months postpartum. If effective, this approach has great potential for scale up where most needed.

ELIGIBILITY:
Inclusion Criteria:

* mothers of healthy infants being discharged from participating maternities who intend to attend well-baby clinic visits in the same health care facilities until the child will be at least 6 months

Exclusion Criteria:

* refusal to participate, not speaking Lingala nor French, unable to breastfeed

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 992 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Early initiation of breastfeeding | Within 1 hour of birth
  initiation of breastfeeding within one hour of birth
Exclusive breastfeeding rate | up to 6 months after birth
  Infants will be classified as exclusively breastfed if they received only breast milk (no water, other liquids, or solids)

SECONDARY OUTCOMES:
Episodes of diarrhea | in the first 6 months of life
Episodes of Lower Respiratory Track Infection | in the first 6 months of life
Partial Breastfeeding rate | up to 6 months after birth
Number of hospitalization | in the first 6 months of life
Number of mothers seeking breastfeeding help | in the first 6 months of life
Amount and type of breastfeeding support given by Health care provider to mothers | in the first 6 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Yotebieng, M.D, MPH, Ph.D, Principal Investigator — University of North Carolina, Chapel Hill; Miriam Labbok, MD, MPH, FACPM, IBCLC, Principal Investigator — University of North Carolina, Chapel Hill; Frieda Behets, Ph.D, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Ksph/Unc-Drc, Kinshasa, Kinshasa, Republic of the Congo

REFERENCES:
- [Result] Yotebieng M, Chalachala JL, Labbok M, Behets F. Infant feeding practices and determinants of poor breastfeeding behavior in Kinshasa, Democratic Republic of Congo: a descriptive study. Int Breastfeed J. 2013 Oct 1;8(1):11. doi: 10.1186/1746-4358-8-11. PMID 24083882
- [Result] Yotebieng M, Labbok M, Soeters HM, Chalachala JL, Lapika B, Vitta BS, Behets F. Ten Steps to Successful Breastfeeding programme to promote early initiation and exclusive breastfeeding in DR Congo: a cluster-randomised controlled trial. Lancet Glob Health. 2015 Sep;3(9):e546-55. doi: 10.1016/S2214-109X(15)00012-1. Epub 2015 Aug 2. PMID 26246225
- [Result] Zivich PN, Kiketa L, Kawende B, Lapika B, Yotebieng M. Vaccination Coverage and Timelines Among Children 0-6 Months in Kinshasa, the Democratic Republic of Congo: A Prospective Cohort Study. Matern Child Health J. 2017 May;21(5):1055-1064. doi: 10.1007/s10995-016-2201-z. PMID 28058663
- [Result] Brazeau NF, Tabala M, Kiketa L, Kayembe D, Chalachala JL, Kawende B, Lapika B, Meshnick SR, Yotebieng M. Exclusive Breastfeeding and Clinical Malaria Risk in 6-Month-Old Infants: A Cross-Sectional Study from Kinshasa, Democratic Republic of the Congo. Am J Trop Med Hyg. 2016 Oct 5;95(4):827-830. doi: 10.4269/ajtmh.16-0011. Epub 2016 Aug 22. PMID 27549632
- [Derived] Agler RA, Zivich PN, Kawende B, Behets F, Yotebieng M. Postpartum depressive symptoms following implementation of the 10 steps to successful breastfeeding program in Kinshasa, Democratic Republic of Congo: A cohort study. PLoS Med. 2021 Jan 11;18(1):e1003465. doi: 10.1371/journal.pmed.1003465. eCollection 2021 Jan. PMID 33428617
- [Derived] Zivich P, Lapika B, Behets F, Yotebieng M. Implementation of Steps 1-9 to Successful Breastfeeding Reduces the Frequency of Mild and Severe Episodes of Diarrhea and Respiratory Tract Infection Among 0-6 Month Infants in Democratic Republic of Congo. Matern Child Health J. 2018 May;22(5):762-771. doi: 10.1007/s10995-018-2446-9. PMID 29417366